CLINICAL TRIAL: NCT02239991
Title: Management of Perioperative Coagulopathy With Thromboelastometry (ROTEM) in Liver Transplant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Luiz Henrique Ide Yamauchi, Physician, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1986-14
Record Dates: First submitted 2014-09-03; First posted 2014-09-15 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Blood Coagulation Disorders; Evidence of Liver Transplantation; Liver Cirrhosis
Keywords: Point of care; perioperative hemostasis; thromboelastometry; bleeding risk; end-stage liver disease; hepatic coagulopathy; whole blood coagulation
MeSH Terms: conditions — Blood Coagulation Disorders; Liver Cirrhosis; End Stage Liver Disease | interventions — Thrombelastography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Historical control (No Intervention): Group of patients that had their coagulopathy secondary to the liver transplant treated based on conventional laboratory tests. Before the implementation of thromboelastometry.
- Intervention (Experimental): Group of cirrhotic bleeding patients that are treated with a bed side, point of care protocol based on thromboelastometry to guide transfusion and manage coagulopathy
  Interventions: Procedure: Thromboelastometry

INTERVENTIONS:
Procedure: Thromboelastometry — Group of cirrhotic bleeding patients that are treated with a bed side, point of care protocol based on thromboelastometry to guide transfusion and manage coagulopathy
  Other Names: point of care bleeding management; ROTEM; viscoelastic test
  Arms: Intervention

SUMMARY:
A point-of-care bleeding management protocol based on global viscoelastic test (thromboelastometry) can change the amount of blood products used during orthotopic liver transplant.

DETAILED DESCRIPTION:
Patients with liver disease frequently acquire a complex disorder of hemostasis secondary to their disease.

The fundamental key to the management of coagulopathy of cirrhotic patient is the knowledge that hepatic dysfunction results in impairment of both pro-hemostatic factors as anti-hemostatic factors in a disproportionate manner which can lead to a clinical picture of both bleeding and thrombosis.

Routine tests of coagulation as prothrombin time (PT, INR) and activated partial thromboplastin time (APTT) although prolonged in cirrhotic patients cannot predict bleeding.

Global viscoelastic test of whole blood (TEG / ROTEM) produce a dynamic composite image of the entire coagulation process and have the potential to provide clinically relevant information in patients with liver disease allowing rational use of blood products during liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* all patients from the national list of liver transplant assigned to have their transplant in Hospital Israelita Albert Einstein who gave free and clarified consent term.

Exclusion Criteria:

* acute liver failure
* age under 18
* combined transplant
* re transplantation less than 30 days
* incomplete medical records, more than 20% of missing data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-08 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Units of packed red blood cells (PRBCs) | intraoperative
  A prospective cohort study based on a point-of care protocol to monitor and manage the coagulopathy based on rotational thromboelastometry (ROTEM) in liver transplant with a historical control. Fifty patients will be managed by ROTEM protocol and will be compared with an equal number of historical controls treated according to the traditional protocol based on clinical and laboratory tests. The aim of this prospective study is to show a reduction in 20% of PRBCs transfusion during liver transplant.

SECONDARY OUTCOMES:
mortality | 30 days
  All patients in interventional group will be followed for a period of 30 days.
Sepsis | During intensive care unit
  Sepsis is defined as the presence (probable or documented) of infection together with systemic manifestations of infection. All patients in interventional group will be followed for a period of 30 days.
Acute respiratory distress syndrome | During intensive care unit
  A chest X-ray will be done in all patients and will be followed for a period of 30 days. A chest X-ray can reveal which parts of your lungs have fluid in them
Mechanical ventilation | During intensive care unit
  All patients in interventional group will be followed for a period of 30 days and will be noted the number of days under mechanical ventilation.
Intensive care unit | up to 30 days
  Length of intensive care unit stay

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Henrique Ide Yamauchi, Physician, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Rana A, Petrowsky H, Hong JC, Agopian VG, Kaldas FM, Farmer D, Yersiz H, Hiatt JR, Busuttil RW. Blood transfusion requirement during liver transplantation is an important risk factor for mortality. J Am Coll Surg. 2013 May;216(5):902-7. doi: 10.1016/j.jamcollsurg.2012.12.047. Epub 2013 Mar 9. PMID 23478547
- [Background] Maxwell MJ, Wilson MJA. Complications of blood transfusion. Continuing Education in Anaesthesia. Crit Care Pain 2006; 6: 225-229
- [Background] Massicotte L, Sassine MP, Lenis S, Roy A. Transfusion predictors in liver transplant. Anesth Analg. 2004 May;98(5):1245-51, table of contents. doi: 10.1213/01.ane.0000111184.21278.07. PMID 15105195
- [Background] Liu LL, Niemann CU. Intraoperative management of liver transplant patients. Transplant Rev (Orlando). 2011 Jul;25(3):124-9. doi: 10.1016/j.trre.2010.10.006. Epub 2011 Apr 21. PMID 21514137
- [Background] Ozier Y, Pessione F, Samain E, Courtois F; French Study Group on Blood Transfusion in Liver Transplantation. Institutional variability in transfusion practice for liver transplantation. Anesth Analg. 2003 Sep;97(3):671-679. doi: 10.1213/01.ANE.0000073354.38695.7C. PMID 12933381
- [Background] de Boer MT, Christensen MC, Asmussen M, van der Hilst CS, Hendriks HG, Slooff MJ, Porte RJ. The impact of intraoperative transfusion of platelets and red blood cells on survival after liver transplantation. Anesth Analg. 2008 Jan;106(1):32-44, table of contents. doi: 10.1213/01.ane.0000289638.26666.ed. PMID 18165548
- [Background] Liu S, Fan J, Wang X, Gong Z, Wang S, Huang L, Xing T, Li T, Peng Z, Sun X. Intraoperative cryoprecipitate transfusion and its association with the incidence of biliary complications after liver transplantation--a retrospective cohort study. PLoS One. 2013 May 10;8(5):e60727. doi: 10.1371/journal.pone.0060727. Print 2013. PMID 23675406 (Retraction: PMID 31491019 PLoS One. 2019 Sep 6;14(9):e0222377)
- [Background] Ramos E, Dalmau A, Sabate A, Lama C, Llado L, Figueras J, Jaurrieta E. Intraoperative red blood cell transfusion in liver transplantation: influence on patient outcome, prediction of requirements, and measures to reduce them. Liver Transpl. 2003 Dec;9(12):1320-7. doi: 10.1016/jlts.2003.50204. PMID 14625833
- [Background] Cacciarelli TV, Keeffe EB, Moore DH, Burns W, Busque S, Concepcion W, So SK, Esquivel CO. Effect of intraoperative blood transfusion on patient outcome in hepatic transplantation. Arch Surg. 1999 Jan;134(1):25-9. doi: 10.1001/archsurg.134.1.25. PMID 9927126
- [Background] Goodnough LT, Brecher ME, Kanter MH, AuBuchon JP. Transfusion medicine. First of two parts--blood transfusion. N Engl J Med. 1999 Feb 11;340(6):438-47. doi: 10.1056/NEJM199902113400606. No abstract available. PMID 9971869
- [Background] Goodnough LT, Brecher ME, Kanter MH, AuBuchon JP. Transfusion medicine. Second of two parts--blood conservation. N Engl J Med. 1999 Feb 18;340(7):525-33. doi: 10.1056/NEJM199902183400706. No abstract available. PMID 10021474
- [Background] Spahn DR, Casutt M. Eliminating blood transfusions: new aspects and perspectives. Anesthesiology. 2000 Jul;93(1):242-55. doi: 10.1097/00000542-200007000-00035. No abstract available. PMID 10861168
- [Background] Weber CF, Gorlinger K, Meininger D, Herrmann E, Bingold T, Moritz A, Cohn LH, Zacharowski K. Point-of-care testing: a prospective, randomized clinical trial of efficacy in coagulopathic cardiac surgery patients. Anesthesiology. 2012 Sep;117(3):531-47. doi: 10.1097/ALN.0b013e318264c644. PMID 22914710
- [Background] Davenport R, Khan S. Management of major trauma haemorrhage: treatment priorities and controversies. Br J Haematol. 2011 Dec;155(5):537-48. doi: 10.1111/j.1365-2141.2011.08885.x. Epub 2011 Oct 21. PMID 22017416
- [Background] Saner FH, Gieseler RK, Akiz H, Canbay A, Gorlinger K. Delicate balance of bleeding and thrombosis in end-stage liver disease and liver transplantation. Digestion. 2013;88(3):135-44. doi: 10.1159/000354400. Epub 2013 Sep 5. PMID 24008288
- [Background] Tripodi A, Salerno F, Chantarangkul V, Clerici M, Cazzaniga M, Primignani M, Mannuccio Mannucci P. Evidence of normal thrombin generation in cirrhosis despite abnormal conventional coagulation tests. Hepatology. 2005 Mar;41(3):553-8. doi: 10.1002/hep.20569. PMID 15726661
- [Background] Kang YG, Martin DJ, Marquez J, Lewis JH, Bontempo FA, Shaw BW Jr, Starzl TE, Winter PM. Intraoperative changes in blood coagulation and thrombelastographic monitoring in liver transplantation. Anesth Analg. 1985 Sep;64(9):888-96. PMID 3896028
- [Background] Trzebicki J, Flakiewicz E, Kosieradzki M, Blaszczyk B, Kolacz M, Jureczko L, Pacholczyk M, Chmura A, Lagiewska B, Lisik W, Wasiak D, Kosson D, Kwiatkowski A, Lazowski T. The use of thromboelastometry in the assessment of hemostasis during orthotopic liver transplantation reduces the demand for blood products. Ann Transplant. 2010 Jul-Sep;15(3):19-24. PMID 20877262
- [Background] Agarwal A, Sharma N, Vij V. Point-of-care coagulation monitoring during liver transplantation. Trends in Anaesth and Crit Care. 2013;3:42-48.
- [Background] Blasi A, Beltran J, Pereira A, Martinez-Palli G, Torrents A, Balust J, Zavala E, Taura P, Garcia-Valdecasas JC. An assessment of thromboelastometry to monitor blood coagulation and guide transfusion support in liver transplantation. Transfusion. 2012 Sep;52(9):1989-98. doi: 10.1111/j.1537-2995.2011.03526.x. Epub 2012 Feb 5. PMID 22304465
- [Background] McCluskey SA, Karkouti K, Wijeysundera DN, Kakizawa K, Ghannam M, Hamdy A, Grant D, Levy G. Derivation of a risk index for the prediction of massive blood transfusion in liver transplantation. Liver Transpl. 2006 Nov;12(11):1584-93. doi: 10.1002/lt.20868. PMID 16952177
- [Background] Ganter MT, Hofer CK. Coagulation monitoring: current techniques and clinical use of viscoelastic point-of-care coagulation devices. Anesth Analg. 2008 May;106(5):1366-75. doi: 10.1213/ane.0b013e318168b367. PMID 18420846
- [Background] Bauters A, Mazoyer E. Apport de la thromboe ́lastome ́trie rotative (ROTEM) pour l'exploration de l'he ́mostase: inte ́reˆt en pratique clinique. Revue francophone des laboratoires 2007; 393: 45-50
- [Background] Luddington RJ. Thrombelastography/thromboelastometry. Clin Lab Haematol. 2005 Apr;27(2):81-90. doi: 10.1111/j.1365-2257.2005.00681.x. PMID 15784122
- [Background] Tanaka KA, Bader SO, Gorlinger K. Novel approaches in management of perioperative coagulopathy. Curr Opin Anaesthesiol. 2014 Feb;27(1):72-80. doi: 10.1097/ACO.0000000000000025. PMID 24263685
- [Background] Tanaka KA, Bolliger D, Vadlamudi R, Nimmo A. Rotational thromboelastometry (ROTEM)-based coagulation management in cardiac surgery and major trauma. J Cardiothorac Vasc Anesth. 2012 Dec;26(6):1083-93. doi: 10.1053/j.jvca.2012.06.015. Epub 2012 Aug 3. No abstract available. PMID 22863406
- [Background] Romero FA, Razonable RR. Infections in liver transplant recipients. World J Hepatol. 2011 Apr 27;3(4):83-92. doi: 10.4254/wjh.v3.i4.83. PMID 21603030